CLINICAL TRIAL: NCT03801551
Title: Validation of a Tool for the Dimensional Assessment of Apathy in a Population Suffering From Schizophrenia.
Acronym: HANDI-AS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Niort (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CH-NIORT-CREHPSY-01-2017
Record Dates: First submitted 2018-12-11; First posted 2019-01-11 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-07

CONDITIONS: Schizophrenia
Keywords: apathy; schizophrenia
MeSH Terms: conditions — Schizophrenia; Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Experimental)
  Interventions: Diagnostic Test: Validate according to psychometric criteria, a dimensional measure of apathy in a population suffering from schizophrenia spectrum disorder and other psychotic disorders (according to DSM-5 criteria).

INTERVENTIONS:
Diagnostic Test: Validate according to psychometric criteria, a dimensional measure of apathy in a population suffering from schizophrenia spectrum disorder and other psychotic disorders (according to DSM-5 criteria). — Validate according to psychometric criteria, a dimensional measure of apathy in a population suffering from schizophrenia spectrum disorder and other psychotic disorders (according to DSM-5 criteria).

SUMMARY:
Schizophrenia affects about 1% of the world's population. According to the WHO, it was one of the ten most worrying pathologies of the twenty-first century. The situation of psychic disability that results impacted the entire life course. This disease is characterized by positive symptoms (delirium, hallucination, psychotic agitation) and negative symptoms and disorganization (destructuring of thought, language and behavior). Cognitive disorders are easily measurable in the spectrum of schizophrenia and are quantifiable with some tools to measure the level of performance of the individual in different areas.

In these patients apathy is found in one out of two cases (prevalence of 51%), so it is a widespread negative symptom. Apathy corresponds to a pathology of voluntary action that can exist in different forms, resulting from the alteration of one or more mechanisms. It is a predictor of functional outcomes, regardless of positive symptoms or depression.

Studies of people with head injuries have found a link between frontal cognitive impairment and apathy. The recognition, the identification of the dimensional mechanisms of apathy and the understanding of the links with cognitive disorders are therefore a major issue in the improvement of the functional prognosis. Moreover, these mechanisms are currently little studied in the spectrum of schizophrenia.

There are currently questionnaires to show the presence or absence of apathy, such as the Apathy Evaluation Scale or the Lille Apathy Rating Scale. However most scales offer a global apathy score and the proposed treatments are limited due to the difficulty in identifying the dimensions and understanding of the underlying mechanisms of their own.

The potentiality of apathy to become a source of disability is now widely recognized. It is therefore important to consider the expression of this handicap in terms of the repercussions that this disorder may have on the daily lives of patients. There are questionnaires to measure the functional autonomy of patients with a psychic disorder. Apathy is also an obstacle to supporting patients in psychiatry.

The lack of knowledge and underestimation of apathy and its mechanisms in schizophrenia, in addition to overworking the psychiatric health sector, favor a drift towards the institutionalization of the person, with its medico-economic consequences on the system.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 55 years old
* According to the DSM-5 criteria: spectrum of schizophrenia and other psychotic disorders (excluding psychotic disorder induced by a substance, drug or other medical condition as well as schizotypal personality disorder) in relation to the medical file and confirmed by the MINI test.
* Stable symptomatology (clinical assessment) during the month prior to inclusion
* Substantive psychotropic treatment unchanged during the month prior to inclusion (25% change).
* Reading and writing in French acquired.
* Persons who received informed information about the study and who co-signed, with the investigator, a consent to participate in the study
* After signing the consent by persons under guardianship, signed consent for participation by the tutor.
* For persons under guardianship, signature of the consent under the curator's assistance.
* Affiliate or Social Security Entitlement

Exclusion Criteria:

* IQ score < 70 (intellectual disability measured by f-NA)
* Neurological disorders of vascular, infectious or neurodegenerative origin, dyschromatopsia.
* Taking somatic drugs with a cerebral or mental impact (eg corticosteroids).
* Resistance to neuroleptics.

Addiction to cannabis, alcohol or other substances (> 2 / week) according to DSM-5 criteria, except tobacco.

* Simultaneous participation in a remediation program targeting neurocognitive deficits.
* Refusal of consent of the person.
* For persons under guardianship: refusal of consent of the legal representative for participation in this study.
* For persons under curatorship: no information of the legal representative for participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
validation of the scale | 1 month
  The DAS is a self-rated multidimensional apathy measure, consisting of 24 items assessing Executive, Initiation and Emotional dimensions of apathy. Each item was rated on a 4-point Likert scale (Hardlyever, Occasionally, Often and Almost always), the minimum score for each subscale is 0 (least apathy) and the maximum 24 (most apathy), with a total score of 72. The French Dimensional Apathy Scale (f-DAS) was firstly tested on healthy participants. The Cronbach Alpha of f-DAS was 0.71 and reflected an acceptable internal reliability.

CONTACTS AND LOCATIONS:
Overall Officials: LISE M'BAREK, Study Director — Centre Hospitalier de Niort - France
Locations (2):
- France (2):
  - Centre Hospitalier Esquirol, Limoges
  - Centre Hospitalier de Niort, Niort